CLINICAL TRIAL: NCT00976794
Title: Efficacy and Tolerability of the Combination of LIthium and CArbamazepine Compared to Lithium and VALproic Acid in the Treatment of Young Bipolar Patients
Brief Title: Efficacy of Combined Treatment for Young Bipolar I Disorder
Acronym: LICAVAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., MD PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2898
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Bipolar I Disorder
Keywords: BD I
MeSH Terms: interventions — Lithium; Carbamazepine; Valproic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lithium plus carbamazepine (Experimental): combination of the two drugs in standard dosage
  Interventions: Drug: lithium plus carbamazepine
- lithium plus valproate (Active Comparator): combination of the two drugs in standard dosage
  Interventions: Drug: lithium plus valproate

INTERVENTIONS:
Drug: lithium plus carbamazepine — Lithium: Starting at 600 mg daily, dose weekly adjusted according to blood serum level (0,6 -1,2mEq/l), efficacy and tolerability.
  Carbamazepine : Starting at 200mg daily and getting 600 mg daily at the end of the first week. Dose weekly adjusted according to blood serum level (8 and 12µg/ml), efficacy and tolerability
  Arms: lithium plus carbamazepine
Drug: lithium plus valproate — Lithium: Starting at 600 mg daily, dose weekly adjusted according to blood serum level (0,6 -1,2mEq/l), efficacy and tolerability.
  Valproic acid: Starting at 500mg daily, dose weekly adjusted according to blood serum level (50 and 125µg/ml), efficacy and tolerability.
  Arms: lithium plus valproate

SUMMARY:
The purpose of this study is to determine the efficacy of the combination of lithium and carbamazepine compared with lithium and valproate treating young bipolar patients.

DETAILED DESCRIPTION:
After the diagnostic assessments, the patients are allocated for one of the following groups of treatment:

Group I: lithium + valproic acid

Group II: lithium + carbamazepine

Patients will be followed up for 8 weeks in phase I (acute treatment), 6 months in phase II (continuation treatment) and 12 months in phase III (maintenance treatment). Scales raters will be blind to the treatment.

During phase II and III will continue only patients that achieve response, measured according to initial symptoms score in phase I.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bipolar Disorder, type I, in current episode (manic/hypomanic, mixed or depression)
* The patient or his (her) legal representative should understand the nature of the study and sign the Informed Consent.

Exclusion Criteria:

* Schizophrenia or schizoaffective disorder
* Mental retardation
* Unstable clinical diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The main outcome will be the number of patients that achieve and remain in remission to each treatment at the end of each phase of the study. | August 2012

SECONDARY OUTCOMES:
Secondary outcome will include the proportion of patients that had response but not remission to each treatment at the end of each phase of the study | August 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry - University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fountoulakis KN, Vieta E, Sanchez-Moreno J, Kaprinis SG, Goikolea JM, Kaprinis GS. Treatment guidelines for bipolar disorder: a critical review. J Affect Disord. 2005 May;86(1):1-10. doi: 10.1016/j.jad.2005.01.004. PMID 15820265
- [Derived] Missio G, Moreno DH, Demetrio FN, Soeiro-de-Souza MG, Dos Santos Fernandes F, Barros VB, Moreno RA. A randomized controlled trial comparing lithium plus valproic acid versus lithium plus carbamazepine in young patients with type 1 bipolar disorder: the LICAVAL study. Trials. 2019 Oct 26;20(1):608. doi: 10.1186/s13063-019-3655-2. PMID 31655626
- [Derived] Campos RN, Costa LF, Bio DS, Soeiro de Souza MG, Garcia CR, Demetrio FN, Moreno DH, Moreno RA. LICAVAL: combination therapy in acute and maintenance treatment of bipolar disorder. Trials. 2010 Jun 23;11:72. doi: 10.1186/1745-6215-11-72. PMID 20573223